CLINICAL TRIAL: NCT05802953
Title: Investigation of the Relationship of Individual, Physical and Psychosocial Characteristics With Quality of Life in Temporomandibular Joint Dysfunction
Brief Title: Quality of Life in Temporomandibular Joint Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2022/5
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Temporomandibular Joint Dysfunction Syndrome; Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Ergonomics; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temporomandibular joint dysfunction group: The group will include patients with temporomandibular joint dysfunction.
  Interventions: Other: Physical assessments; Other: Questionnaire

INTERVENTIONS:
Other: Physical assessments — Physical assessments include the presence of joint sounds (yes/no), Fonseca Anamnestic Questionnaire, tenderness/pressure pain threshold rating, muscle strengths assessments, temporomandibular joint and cervical region range of motion measurements, and pain.
Other: Questionnaire — General Health Questionnaire-28 and SF-36 will be apply.

SUMMARY:
It is planned to examine the relationship between quality of life in patients with temporomandibular joint dysfunction and the patient's individual, physical and psychosocial characteristics.

DETAILED DESCRIPTION:
A recent study showed that individuals with TMD have a lower quality of life than healthy controls. In addition, it was determined in the study that investigating the quality of life is insufficient. Future studies should search for psychosocial aspects related to TMD. The aim of this study is to individual the physical and psychosocial characteristics of individuals with Axis I TMD and examine their relationship with quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being in group I according to RDC/TMD Axis I,

Exclusion Criteria:

* Any treatment for temporomandibular joint dysfunction (TMD) in the last six months
* Having dental problems
* Having any disorder and/or disease involving structures and/or masticatory muscles associated with TMD
* Having a history of trauma in the head and neck region,
* Having previously undergone temporomandibular joint surgery,
* Using corticosteroid and anticonvulsant drugs
* Patients who have received physiotherapy and rehabilitation related to the temporomandibular joint in the last six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be conducted in Afyonkarahisar Health Science University Faculty of Dentistry. 18-85 aged patients with TMD will be included.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores | 10 minutes
  The quality of life will be assess using SF-36. This questionnaire has 8 sections and 36 items. The sections evaluate health between 0-100 and the higher the score indicates the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided